CLINICAL TRIAL: NCT02591407
Title: A Prospective Randomized Clinical Trial Comparing the Transversus Abdominis Plane Block (TAP) Versus Epidural Anesthesia For Enhanced Recovery Pathway Perioperative Management of Pain in Elective Colorectal Surgery
Brief Title: Trial Comparing Transversus Abdominis Plane Block Versus Epidural Anesthesia for Pain Management in Colorectal Surgery
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Principal Investigator, Robert K Cleary, Colon and Rectal Surgeon, Trinity Health Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR 15-1618
Record Dates: First submitted 2015-10-07; First posted 2015-10-29 (Estimated); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Rectal Cancer; Colonic Diverticulosis
Keywords: Continuous Epidural Analgesia; Transversus Abdominis Plane block
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulosis, Colonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP Block- Exparel (Active Comparator): Transversus abdominis plane block utilizing the medication Exparel®
  Interventions: Procedure: TAP Block
- Continuous Epidural Analgesia (Active Comparator): Continuous Epidural Analgesia
  Interventions: Procedure: Continuous Epidural Analgesia

INTERVENTIONS:
Procedure: TAP Block — This is a one time injection of Exparel in the plane between the internal oblique and transversus abdominis muscles
  Other Names: Exparel
  Arms: TAP Block- Exparel
Procedure: Continuous Epidural Analgesia — Epidural catheter placed prior to the operation in the standard fashion
  Arms: Continuous Epidural Analgesia

SUMMARY:
The primary outcome for this study is the Numeric Pain Score (NPS) for elective patients undergoing elective colorectal surgery that have been randomized to transversus abdominis plane block or epidural anesthesia for the management of perioperative pain in elective colorectal surgery.

DETAILED DESCRIPTION:
Adequate peri-operative analgesia is a vital component of post-operative management for patients undergoing colon and rectal surgery, affecting hospital length of stay, quality of life, and patient outcomes. There are many options for the peri-operative management of pain after elective colorectal surgery.

This is a randomized clinical trial comparing the transversus abdominis plane block using Exparel® to epidural anesthesia for the enhanced recovery pathway perioperative management of pain for elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open and minimally invasive (laparoscopic and robotic) colon and rectal surgery for colorectal neoplasia, diverticulitis, and other diseases of the colon and rectum;
* Surgical procedure either through standard open or minimal invasive approach (laparoscopic or robotic);
* Patients > 18 years of age;
* Able to provide informed written consent
* Patients capable of completing questionnaires at the time of consent

Exclusion Criteria:

* Documented allergic reaction to morphine, hydromorphone, lidocaine, bupivicaine and/or fentanyl;
* Contra-indication to placement of epidural catheter (spinal stenosis, spinal fusion, elevated International Normalized Ratio (INR), anticoagulation, patient refusal, etc) or TAP block (patient refusal);
* Urgent or emergent surgery precluding epidural catheter placement or TAP block;
* Systemic Infection contraindicating epidural catheter placement or TAP block;
* Unwillingness to participate in follow up assessments;
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Cleary, MD, Principal Investigator — Saint Joseph Mercy Hospital
Locations (1):
- Saint Joseph Mercy Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felling DR, Jackson MW, Ferraro J, Battaglia MA, Albright JJ, Wu J, Genord CK, Brockhaus KK, Bhave RA, McClure AM, Shanker BA, Cleary RK. Liposomal Bupivacaine Transversus Abdominis Plane Block Versus Epidural Analgesia in a Colon and Rectal Surgery Enhanced Recovery Pathway: A Randomized Clinical Trial. Dis Colon Rectum. 2018 Oct;61(10):1196-1204. doi: 10.1097/DCR.0000000000001211. PMID 30192328
- See also: American Society of Colon and Rectal Surgeons — http://www.fascrs.org

RESULTS

PARTICIPANT FLOW:
Period: Randomization
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Started | 101 | 99
Completed | 89 | 94
Not Completed | 12 | 5
Not completed — Cancelled surgery | 5 | 3
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Emergency surgery | 0 | 1
Period: Follow-up
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Started | 89 | 94
Completed | 87 | 92
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 2
Period: Analysis
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Started | 87 | 92
Completed | 87 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block- Exparel | Continuous Epidural Analgesia | Total
Number analyzed (Participants) | 92 | 87 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] — age, at consent (years)
  years | 62.05 (11.79) | 62.06 (11.12) | 62.05 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 76
  Male | 50 | 53 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 6 | 8 | 14
  White | 85 | 77 | 162
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 92 | 87 | 179
Tobacco use [Count of Participants; unit: Participants] | 12 | 15 | 27
Alcohol use [Count of Participants; unit: Participants] | 1 | 2 | 3
Steroids use [Count of Participants; unit: Participants] | 2 | 2 | 4
Opioid use [Count of Participants; unit: Participants] | 1 | 1 | 2
Hypertension [Count of Participants; unit: Participants] | 51 | 48 | 99
Coronary artery disease [Count of Participants; unit: Participants] | 11 | 8 | 19
Congestive heart failure [Count of Participants; unit: Participants] | 5 | 4 | 9
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 4 | 3 | 7
Sleep apnea [Count of Participants; unit: Participants] | 8 | 7 | 15
Diabetes mellitus [Count of Participants; unit: Participants] | 13 | 15 | 28
Renal disease [Count of Participants; unit: Participants] | 2 | 5 | 7
Deep Vein Thrombosis/Pulmonary Embolism (DVT/PE) [Count of Participants; unit: Participants] | 8 | 1 | 9
Disseminated cancer [Count of Participants; unit: Participants] | 5 | 5 | 10
Previous abdominal surgery [Count of Participants; unit: Participants] | 41 | 30 | 71

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Mean Numeric Pain Scale.
Description: Measured by patient completing the Numeric Pain Scale (NPS) on post-operative day 0,1,2,3. Numeric Pain Scale is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
  Data from all the specified time points above (post-operative day 0,1,2,3) was averaged into a single value.
Time Frame: Post-operative day 0,1,2,3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
units on a scale | 2.12 (1.44) | 2.32 (1.44)

2. Primary Outcome: Overall Benefits of Analgesia Score (OBAS)
Description: Measured by the patient completing the OBAS survey on postoperative days 0,1,2,3. The OBAS is a multi-dimensional quality assessment instrument to measure patients' benefit from postoperative pain therapy.
  1. Rate your current pain at rest on a scale between 0=minimal pain and 4=maximum imaginable pain 2-6. Grade any distress and bother from vomiting in the past 24 h (0=not at all to 4=very much: same scale for remaining Qs about itching, sweating, freezing, dizziness on the scale).
  7. Rate your satisfaction with your pain treatment on a scale between 0=not at all and 4= very much
  To calculate the OBAS score, compute the sum of scores in items 1-6 and add the '4-(score in item 7)'. The range of scores is from 0 (best) to 28 (worst).
  Data from all the specified time points above (post-operative day 0,1,2,3) was averaged into a single value.
Time Frame: Post-operative day 0,1,2,3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
units on a scale | 0.48 (0.52) | 0.37 (0.31)

3. Secondary Outcome: Patient Use of Narcotic Analgesia Post-op Day 0
Description: Patient use of narcotic analgesia post-operative day 0 including Fentanyl from epidural
Time Frame: Post-operative day 0
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
Morphine milligram equivalents | 80.20 [58.41 to 110.12] | 54.64 [50.35 to 59.31]

4. Secondary Outcome: Patient Use of Narcotic Analgesia Post-operative Day 0
Description: Patient use of narcotic analgesia post operative day 0 excluding Fentanyl from epidural.
Time Frame: Post-operative day 0
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
Morphine milligram equivalents | 27.55 [20.77 to 36.55] | 54.64 [50.35 to 59.31]

5. Secondary Outcome: Patient Use of Narcotic Analgesia Post-operative Day 3
Description: Patient use of narcotic analgesia post-operative day 3 including Fentanyl from epidural
Time Frame: Post-operative day 3
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
Morphine milligram equivalents | 0.34 [0.15 to 0.77] | 0.22 [0.10 to 0.45]

6. Secondary Outcome: Patient Use of Narcotic Analgesia Post-operative Day 1
Description: Patient use of narcotic analgesia post operative day 1 including Fentanyl from epidural
Time Frame: Post-operative day 1
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
Morphine milligram equivalents | 71 [53.42 to 94.36] | 13.34 [8.14 to 21.86]

7. Secondary Outcome: Patient Use of Narcotic Analgesia Post-operative Day 2
Description: Patient use of narcotic analgesia post operative day 2 including Fentanyl from epidural
Time Frame: Post-operative day 2
Measure: Mean (Full Range); unit: Morphine milligram equivalents
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
Number analyzed (Participants) | 87 | 92
Morphine milligram equivalents | 3.11 [1.52 to 6.38] | 2.61 [1.33 to 5.14]

ADVERSE EVENTS:
Time Frame: 6 months from treatment.
Arm/Group | Continuous Epidural Analgesia | TAP Block- Exparel
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/92
Other Adverse Events (participants affected / at risk) | 0/87 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT02591407/Prot_SAP_000.pdf